CLINICAL TRIAL: NCT00437814
Title: Effect of Ketamine (Ketalar) on Intracranial Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KETICP.CTIL
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Traumatic Brain Injury; Intracranial Hypertension
Keywords: Ketamine; Traumatic Brain Injury; Intracranial Hypertension
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension | interventions — Ketamine

INTERVENTIONS:
Drug: Ketamine, effect on intracranial pressure

SUMMARY:
Objectives: Ketamine is an effective, short-acting anesthetic drug, which does not decrease blood pressure. It is widely stated that Ketamine increases intracranial pressure (ICP), which prevents its use in many emergency situations, specifically in patients with traumatic brain injury (TBI) and with increased ICP. Based on previous clinical experience, we hypothesized that Ketamine decreases - rather than increases - ICP.

Methods: Prospective, controlled, clinical trial. Children with ICP monitoring will receive a single Ketamine dose (1-1.5 mg/kg) either for increased ICP and/or before a potentially distressing activity. Hemodynamic variables, ICP and cerebral perfusion pressure (CPP) will be recorded 1 minute before and every minute for 10 minutes following Ketamine administration (Before/after design).

DETAILED DESCRIPTION:
Objectives: Ketamine is an effective, safe, rapid, short-acting anesthetic drug, and - contrary to all other anesthetic drugs - it does not decrease blood pressure. It is widely believed that Ketamine increases intracranial pressure (ICP), which prevents its use in many emergency situations, including trauma and specifically in patients with traumatic brain injury (TBI) and with increased ICP. Based on our previous clinical experience in patients with ICP monitoring, Ketamine did not increase ICP. We therefore hypothesize that Ketamine decreases - rather than increases - ICP.

Methods: Prospective, controlled, clinical trial performed in a Pediatric ICU of a regional trauma center. Children with ICP monitoring receive a single Ketamine dose (1-1.5 mg/kg) either for increased ICP and/or before a potentially distressing activity. Hemodynamic variables, ICP and cerebral perfusion pressure (CPP) will be recorded 1 minute before and every minute for 10 minutes following Ketamine administration (before/after study design).

Parents/guardian of patients will be informed and asked to sign an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Children who have an ICP monitoring device, who either have increased ICP and/or who should undergo a potentially distressing activity (suction, position change etc.).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2007-02

PRIMARY OUTCOMES:
Effect on intracranial pressure
Effect on hemodynamic variables
Effect on cerebral perfusion pressure

CONTACTS AND LOCATIONS:
Overall Officials: Gad Bar-Joseph, MD, Study Director — Director, Pediatric ICU, Rambam Medical Center
Locations (1):
- Pediatric ICU, Rambam Medical Center, Haifa, Israel